CLINICAL TRIAL: NCT03818945
Title: Clinical Efficacy of Giomer Versus Sodium Fluoride Varnish for Management of Hypersensitivity: Randomized Control Trail
Brief Title: the Efficacy of Giomer Versus Sodium Fluoride in the Treatment of Hypersensitivity
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nourane Yasser Ali, Principal investigator in Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Nourane Yasser
Record Dates: First submitted 2019-01-24; First posted 2019-01-28 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Tooth Hypersensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Bifluorid 12

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium Fluoride Varnish (Other)
  Interventions: Drug: Sodium fluoride varnish
- PRG barrier Giomer (Active Comparator)
  Interventions: Drug: shofu PRG barrier coat

INTERVENTIONS:
Drug: shofu PRG barrier coat — Trilaminar structure which forms a type of stable glass ionomer allowing ion release and recharge, while protecting the glass core from the damaging effects of moisture, greatly improving long-term durability.(Na, BO3, Al, SiO3, F,Sr)
  Other Names: Light cured giomer
  Arms: PRG barrier Giomer
Drug: Sodium fluoride varnish — 5% sodium fluoride [22,600 ppm F-]
  Other Names: Biofluoride 5% Fluoride varnish single use dose - Vocoo
  Arms: Sodium Fluoride Varnish

SUMMARY:
to solve the problem of hypersensitivity, I will use two different materials ( Giomer versus Sodium Fluoride) and compare between their effects in reliving the symptoms

DETAILED DESCRIPTION:
The dentin hypersensitivity is characterized by short, sharp pain which can be detected by several methods. The problem is very annoying for the patients and making them seek for effective rapid treatment.

It can affect several teeth in one area of the mouth or only one specific tooth. Careful diagnosis of such condition necessitates precise differentiation of its signs and symptoms from the other causes of tooth sensitivity which may be resulted from dental caries, micro leakage, cracked tooth or fractured restoration. There are two well-known ways to reduce the discomfort of the hypersensitivity either by blocking the exposed dentinal tubules by occluding materials or use some depolarizing agents that reducing the excitability of the intra dental nerves.Most of the desensitizing agents reduces the dentin hypersensitivity by its own way and each one has different long lasting effect. But there are some drawbacks that appeared with their use. Fluoride based agents were appeared in 90's but it was clarified that their high concentration irritated the odontoblasts. Furthermore, the oxalates and potassium nitrate were introduced to treat the hypersensitivity effectively but their effects did not persist for a long period of time.

Sodium fluoride varnish is one from the most commonly used desensitizing agent and its efficacy was approved in many studies. The Giomer varnish containing surface pre-reactive glass particles (S-PRG) is a light-cured protective varnish and it was introduced to promote prolonged protection for the hypersensitive dentin.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 18 to 40 years.
* No gender restriction.
* Patients should have pain score in the visual analog scale two or more.
* Patients must have at least one sensitive tooth in one of four quadrants.

Exclusion Criteria:

* Patients with active carious lesions.
* Needing restorative treatment.
* Receiving periodontal treatment.
* Taking desensitizing treatment in the last 6 months.
* Taking anti-inflammatory drugs.
* Pregnant patients.
* Smokers.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2019-06-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
relieving of hypersensitivity | one month
  The sensitive teeth will be assessed by two stimuli: tactile and thermal stimuli than scored according to the visual analog scale from zero to ten.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Giza, Egypt